CLINICAL TRIAL: NCT06231693
Title: Trastuzumab-deruxtecan in Patients With Triple-negative Metastatic HER2-Low Breast Cancer: Real-world Experience in Brazil
Status: Terminated | Type: Observational
Why Stopped: The study was stopped due to a realignment of strategic priorities
Sponsor: AstraZeneca (Industry)
Collaborators: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Other Study IDs: D9673R00036; 74911423.1.1001.0071 (Other: Hospital Israelita Albert Einstein)
Record Dates: First submitted 2024-01-11; First posted 2024-01-30 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Trastuzumab-deruxtecan
  Interventions: Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — Patients with RE<10% and HER2-Low breast cancer that have received Trastuzumab-deruxtecan in the metastatic setting

SUMMARY:
A national, multicenter, retrospective, observational study (Real-World Evidence-RWE) aimed to assess the efficacy of Trastuzumab-deruxtecan (T-DXd) in patients with triple-negative (RE<10%) metastatic HER2-Low breast cancer.

DETAILED DESCRIPTION:
Data from study DESTINY-04 have established T-DXd as the standard second-line treatment for HER2-Low breast tumors. In that study, about 90% of the population had estrogen-positive receptor (ER+) tumors, under-representing negative ER population. The investigators propose to assess T-DXd efficacy in HER2-Low/ER ≤10% patients in Brazilian population by means of a RWE analysis. Endpoints will be assessment of time to the next treatment, objective response rate, and real-world progression-free survival and real-world overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 18 years old;
* Have advanced, hormone receptor negative (ER ≤10%), HER2-Low (1+ or 2+/FISH negative) breast cancer;
* Have been treated with at least one trastuzumab-deruxtecan dose for advanced disease (incurable) as a second or later line;
* Do not have active CNS metastatic lesions, characterized as stable, asymptomatic lesions and with no targeted treatment for at least 6 months.

Exclusion Criteria:

* Have been previously treated with trastuzumab-deruxtecan (neoadjuvant, adjuvant, other neoplasms);
* Have other active neoplasms (except from non-melanoma skin tumors);
* Have serious or active non-oncology lung diseases;
* Have other primary and concurrent breast tumor with differing receptor profiles.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, with metastatic HER2-Low/ER ≤10% breast tumors, from Brazilian population, who were given TDXd as per usual prescription from their physician
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Time to Next Treatment | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Response Rate | Through study completion, an average of 18 months
Real World Progression Free Survival | Through study completion, an average of 18 months
Real World Overall Survival | Through study completion, an average of 18 months
Epidemiological Features | Through study completion, an average of 18 months
  Age, comorbidities, somatic mutations, pattern of HER2 testing.

CONTACTS AND LOCATIONS:
Overall Officials: Italo Fernandes, MD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (2):
- Brazil (2):
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR_Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9673R00036&attachmentIdentifier=3ed6c586-cf27-4061-9152-2ee459bd2eae&fileName=CSR_Synopsis_Redacted.pdf&versionIdentifier=